CLINICAL TRIAL: NCT00985738
Title: A Randomized Placebo-Controlled Double-Blind Clinical Trial to Assess the Role of Dutasteride in Patients Undergoing 3D Mapping Biopsy in Early Stage Prostate Cancer
Brief Title: Role of Dutasteride in Patients Undergoing 3D Mapping Biopsy in Early Stage Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of Colorado, Denver (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-0247.cc
Record Dates: First submitted 2009-09-11; First posted 2009-09-28 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Early Stage Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dutasteride (Experimental): The drug, Dutasteride, will be administered at 0.5 mg dose and given everyday (QD), for 3 months.
  Interventions: Drug: Dutasteride
- Placebo (Placebo Comparator): The placebo group will receive a placebo drug for 3 months, instead of the intervention drug, Dutasteride.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dutasteride — Dutasteride will be administered at 0.5 mg dose and it will be given every day (QD), for approximately 3 months, followed by 3D mapping biopsy.
  Other Names: Avodart
  Arms: Dutasteride
Other: Placebo — The placebo group will receive the same standard of care as the intervention group, but instead of receiving the intervention drug, Dutasteride, participants will receive a placebo drug for the same 3 month period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of short-term intake of daily Dutasteride in patients with prostate cancer.

DETAILED DESCRIPTION:
This is a study of men who have undergone a standard 10 or more core biopsy for detection of prostate cancer and determined to have prostate cancer by having a Gleason score ≤ 7 (low to moderate risk 2-7). Of these men, one arm of a two arm randomized group will be administered a treatment regime of Dutasteride versus the control group who receive standard of care, prior to mapping biopsy. This proposal aims at studying the apparent effect of the use of Dutasteride (3 months) on initial tumor volume (at diagnosis) in men with low volume cancer before undergoing 3D mapping biopsy.

ELIGIBILITY:
Inclusion Criteria:

* 40-85 year old males
* Patient is newly diagnosed with clinical Stage T1a-T2c prostate cancer based on transrectal guided extended prostate biopsy of at least 10 cores.
* Patient elects to undergo 3D mapping biopsy at our center as part of prostate cancer management.
* Patient will read, understand and sign the informed consent agreement
* Patients must have a life expectancy of at least one year.
* Gleason score ≤ 7 (low to moderate risk 2-7) 7= 3+4
* Percentage positive core rate < 50% based on sextant or extended biopsy technique.
* Prostate Volume (PV) >15 grams.
* Negative imaging studies ( if available) during the staging period such as Bone scan, MRI and CT scan if PSA> 10 ng.dl before initiation of the study drug

Exclusion Criteria:

* Any 5α-reductase inhibitors medications within the past 12 months before enrollment.
* Known hypersensitivity to dutasteride, or other 5α-reductase inhibitors.
* Anticipated blood donation within the next 90 days.
* Serum PSA levels of >20ng/dl.
* Clinical evidence of metastatic prostate cancer.
* Two documented urinary tract infections in the past year
* CHF, MI (within 6 months) or other symptomatic CVS disease
* Other serious diseases (hematological, hepatic, renal, respiratory or psychiatric)
* Enrollment in other studies for any disease in the past 30 days
* Significant urinary incontinence
* Diagnosis of cancer that in not considered cured, except BCC of skin
* Prior transurethral resection of the prostate with a large tissue defect.
* History of abdominoperineal resection for rectal cancer, rectal stenosis, or other major rectal pathology
* Previous or concurrent radiotherapy, hormonal therapy or chemotherapy

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al Barqawi, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The link above provides detail about the Primary Investigator (PI- Al Barqawi MD FRCS) and his research on prostate cancer. In addition, this website includes the PI's resume and publications. — http://www.alprostate.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2009 and 2011, 16 patients were enrolled in the study from the Urologic Oncology clinic and Outpatient Urology clinic.
Pre-assignment Details: Subjects who qualified for the study based on the eligibility criteria were randomized to a placebo or treatment arm. After approximately 90 days (± 10 days), patients returned to undergo 3D mapping biopsy as part of their management of prostate cancer and received the tests/procedures outlined in the study calendar.
Groups:
- Dutasteride: Dutasteride (Avodart) was administered at 0.5 mg dose and was given every day (QD) for 3 months, followed by 3D mapping biopsy.
- Placebo: This group received a placebo followed by 3D mapping biopsy.
Period: Overall Study
Arm/Group | Dutasteride | Placebo
Started | 8 | 8
Completed | 0 | 0
Not Completed | 8 | 8
Not completed — Study closed prematurely | 8 | 8

BASELINE CHARACTERISTICS:
Population: A one sided test of proportions with an alpha level of 0.025 was performed for a conservative Fisher's exact method. It was estimated that an 80% power in a test of proportions with 100 men in each arm would detect a 17% difference in proportion of men with increased tumor volume (upstaging) between the treatment arm and the control arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (6.0) | 65.8 (6.3) | 64.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Effect of Short-term Intake of Daily Dutasteride Prostate Cancer Volume, Distribution Within the Gland and Gleason Score Sum in Patients in Comparison to Placebo After Adjusting for Changes in Prostate Gland Volume.
Description: The effect of Dutasteride intake on the following parameters as detected by mapping biopsy vs. initial trans-rectal biopsy in the treatment arm and the control group: change in prostate gland volume, change in distribution within the gland, and change in Gleason score sum.
Time Frame: 24 Months
Population: "The study was terminated. Study end points were not reached. No data were collected
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 27 months.
Description: Adverse events were monitored throughout the course of the study and 3-months as a follow up period.
Arm/Group | Dutasteride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
This study was terminated due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No